CLINICAL TRIAL: NCT06852417
Title: Health Qigong Alleviates Depressive Symptoms in Older Adults Through Enhanced Executive Attention: a Randomized Controlled Trial
Brief Title: Qigong and Executive Attention in Older Adults with Depressive Symptoms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, LU Yiqing Erin, Research Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15612625
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Intervention; Waitlist Control
Keywords: Health qigong; Baduanjin; executive attention; depressive symptoms
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Baduanjin (Experimental): This arm is for intervention group who will receive health qigong training.
  Interventions: Behavioral: Health qigong training
- Waitlist control (No Intervention): The arm is for control group who will not receive any training.

INTERVENTIONS:
Behavioral: Health qigong training — Participants will receive two 60-minute Baduanjin qigong training sessions every week under the instruction and supervision of qualified qigong instructors over 12 weeks (i.e., 24 sessions in total). Baduanjin qigong consists of eight forms of gentle movements, and it takes about 10 to 15 minutes to complete a full cycle. Participants will learn to practice each form gradually over the first 12 sessions. In the remaining 12 sessions, the participants will go through all the movements 2-3 times, with guided practice on rhythmic breathing and mind regulation (attention to body and breathing) to be performed in coordination with the movements. Instructions on each movement, voice-guide audios, and demonstration videos will be provided for participants' daily self-practice. They will be advised to practice Baduanjin for at least 10 minutes every day.
  Arms: Baduanjin

SUMMARY:
The goal of this randomized controlled trial is to test whether executive attention unpacks the antidepressant effect of Baduanjin (a form of health qigong) in older adults.

The main questions it aims to answer are:

* Is Baduanjin an effective treatment to enhance executive attention in older adults with depressive symptoms?
* Does Baduanjin work through enhanced executive attention to alleviate depressive symptoms in older adults? Researchers will compare Baduanjin with waitlist control. Participants will receive 12-week Baduanjin training (two sessions per week and 60 min per session).

DETAILED DESCRIPTION:
Baduanjin is a type of health qigong that has been shown to effectively reduce depressive symptoms in older adults. However, the cognitive mechanism that explains such antidepressant effect remains unclear. Executive attention represents the cognitive processing that deals with interference and conflict, and it is likely to be a mechanism to unpack Baduanjin's treatment effect on depressive symptoms. There is also a lack of understanding of Badunajin's effects on brain activation in depressed older adults. To address these knowledge gaps, we propose a fully powered randomized controlled trial (RCT) with 198 older adults with at least mild depressive symptoms. They will be randomly assigned to either the active intervention group (12-week Baduanjin training) or the waitlist control group. The primary outcome is executive attention. Secondary outcomes include depressive symptoms, amplitudes of N2 and P3 components (i.e., components of event-related potentials in brain) during attention tasks, and alerting and orienting networks of attention. These outcomes will be assessed at baseline and post-intervention (12 weeks after baseline). Repeated measures ANOVA will be used to test for treatment effects on the primary outcome. Executive attention's mediation effect on the linkage between group (intervention vs waitlist control) and depressive symptoms will be tested with SPSS Macro PROCESS. The Baduanjin-related enhancement in N2 amplitude, P3 amplitude, alerting, and orienting will be explored with repeated measures ANOVA, respectively. Correlation analyses will be used to evaluate the association (i) between changes in N2 and P3 amplitudes and changes in executive attention and (ii) between changes in N2 and P3 amplitudes and changes in depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* have mild or severer levels of depressive symptoms, as indicated by Geriatric Depression Scale scores of 5 or above or Depression Anxiety and Stress Scale-21 depression subscale scores of 4 or above
* self-identified as physically stable and without life-threatening diseases
* be able to communicate in Cantonese or Mandarin.

Exclusion Criteria:

* (have a history of practicing or receiving training in any form of mind-body or regular exercises (including tai chi, yoga, and qigong or regular physical activity > 3 times/week) during the month prior to recruitment
* have changed medications or the dose of medications prescribed for their health condition in the month prior to study enrollment
* have a severe cognitive or language impairment, as indicated by a score of less than 21 on the Montreal Cognitive Assessment
* receiving pharmacological treatment, electroconvulsive therapy, psychotherapy, or psychoeducation for any psychological or psychiatric condition upon the time of recruitment
* be unable to demonstrate satisfactory standing balance.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Executive attention | Baseline and post-intervention (12 weeks after baseline)
  The Attention Network Test (ANT) will be used to assess executive attention. The ANT is a computer-based test based on a combination of Posner's cueing task and the Flanker task. Executive attention will be operationalized as the difference in reaction time (measured in ms) in congruent and incongruent trials.

SECONDARY OUTCOMES:
Depressive symptoms | Baseline and post-intervention (12 weeks after baseline)
  The 8-item Patient Health Questionnaire (PHQ) will be used to assess depressive symptoms. It includes eight items assessing the frequency of depressive symptoms over the previous two weeks on a 4-point scale (0 = never, 3 = almost every day). The total score ranges from 0 to 24, with a higher score indicating a greater severity of depressive symptoms.
Amplitude of N2 component | Baseline and post-intervention (12 weeks after baseline)
  Participants' neurophysiological activity during The Attention Network Test (ANT) will be recorded with a dry electroencephalography (EEG) device, DSI-24 with 21 electrodes. N2 amplitude will be calculated by averaging the amplitudes recorded at the selected electrodes and time windows (210-350 ms).
Amplitude of P3 component | Baseline and post-intervention (12 weeks after baseline)
  Participants' neurophysiological activity during The Attention Network Test (ANT) will be recorded with a dry electroencephalography (EEG) device, DSI-24 with 21 electrodes. P3 amplitude will be calculated by averaging the amplitudes recorded at the selected electrodes and time windows (350-550 ms).
Alerting | Baseline and post-intervention (12 weeks after baseline)
  The Attention Network Test (ANT) will be used to assess alerting. The ANT is a computer-based test based on a combination of Posner's cueing task and the Flanker task. Alerting will be operationalized as the difference in reaction time in no cue trials and center cue trials.
Orienting | Baseline and post-intervention (12 weeks after baseline)
  The Attention Network Test (ANT) will be used to assess orienting. The ANT is a computer-based test based on a combination of Posner's cueing task and the Flanker task. Orienting will be operationalized as the difference in reaction time in center cue trials and spatial cue trials.